CLINICAL TRIAL: NCT01296334
Title: Analgesic and Antihyperalgesic Effects of Morphine and Buprenorphine Following an Experimental Inflammatory Injury in Volunteers.
Brief Title: Analgesic and Antihyperalgesic Effects of Morphine and Buprenorphine
Acronym: PASORII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: mads u werner (Other)
Collaborators: Norpharma A/S (Industry)
Responsible Party: Sponsor-Investigator, mads u werner, MD, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: H-2-2010-115; 2010-022903-23 (EudraCT Number)
Record Dates: First submitted 2011-02-14; First posted 2011-02-15 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Pain
Keywords: opioids; analgesia; secondary hyperalgesia; quantitative sensory testing; inflammatory injury
MeSH Terms: conditions — Pain; Agnosia; Hyperalgesia | interventions — Buprenorphine; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- morphine low dose (Experimental): morphine infusion 10 mg over a 210 min period
  Interventions: Drug: morphine LO
- morphine high dose (Experimental): morphine infusion 20 mg over a 210 min period
  Interventions: Drug: Morphine Hi
- buprenorphine low dose (Experimental): buprenorphine infusion 0.3 mg over a 210 min period
  Interventions: Drug: Buprenorphine LO
- buprenorphine high dose (Experimental): buprenorphine infusion 0.6 mg over a 210 min period
  Interventions: Drug: Buprenorphine Hi
- placebo (Placebo Comparator): placebo (normal saline) infusion 0.6 mg over a 210 min period
  Interventions: Other: saline

INTERVENTIONS:
Drug: morphine LO — intravenous infusion, 10 mg, once, 4 hours
  Other Names: Morfin SAD
  Arms: morphine low dose
Drug: Morphine Hi — intravenous infusion, 20 mg, once, 4 hours
  Other Names: Morfin SAD
  Arms: morphine high dose
Drug: Buprenorphine LO — intravenous infusion, 0.3 mg, once, 4 hours
  Other Names: Temgesic
  Arms: buprenorphine low dose
Drug: Buprenorphine Hi — intravenous infusion, 0.6 mg, once, 4 hours
  Other Names: Temgesic
  Arms: buprenorphine high dose
Other: saline — intravenous infusion, 0.9% saline, once, 4 hours
  Other Names: 0.9% NaCl
  Arms: placebo

SUMMARY:
Tissue injury is associated with pain from the injured site (primary hyperalgesia) and pain from non-injured tissue in the vicinity of the trauma (secondary hyperalgesia). In the present study we investigate primary and secondary hyperalgesia in healthy volunteers following an experimental first degree burn injury.

The objectives are:

* to compare analgesic and anti-hyperalgesic effects of two opioids (morphine and buprenorphine).
* to investigate if these effects are related to the volunteers individual pain sensitivity

DETAILED DESCRIPTION:
Please refer to:

Ravn P, Secher EL, Skram U, Therkildsen T, Christrup LL, Werner MU (2013) Morphine- and buprenorphine-induced analgesia and antihyperalgesia in a human inflammatory pain model: a double-blind, randomized, placebo-controlled, five-arm crossover study. J Pain Res 6: 23-38. 10.2147/JPR.S36827 [doi];jpr-6-023 [pii].

ELIGIBILITY:
Inclusion Criteria:

* healthy individuals
* adequate psychomotor performance to perform pain tests
* pain-sensitive or pain-nonsensitive according to prespecified criteria

Exclusion Criteria:

* known allergy to morphine or buprenorphine
* prior adverse experiences with opioids
* history of abuse
* females not taking P-pills
* skin lesions on the test-sites
* suffering from chronic pain
* medication with analgesics
* BMI > 28
* smoker

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2011-02; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Analgesic and antihyperalgesic effects | 0 to 180 min after a first degree burn injury
  Analgesic effect is assessed by change in primary hyperalgesia (pain rating [VAS]) Antihyperalgesic effect is assessed by reduction in area of hyperalgesia (sq. cm) VAS-area under curve is calculated for 0, 60, 120 and 180 min after first degree burn injury

SECONDARY OUTCOMES:
Difference in analgesic/antihyperalgesic profile between pain-sensitive and pain-non-sensitive individuals | 0-180 min after first degree burn injury
  The ratios between areas under curve (0-180 min after first degree burn injury) for analgesic effect assessed by change in primary hyperalgesia (pain rating VAS])and antihyperalgesic effect assessed by reduction in area of hyperalgesia (sq. cm).

CONTACTS AND LOCATIONS:
Overall Officials: Mads U Werner, MD, DMSc, Study Director — Multidisciplinary Pain Centre 7612, Rigshospitalet, Blegdamsvej 9, DK 2100 Copenhagen O; Lona L Christrup, MSc, PhD, Study Chair — Pharmaceutical Faculty, Copenhagen University
Locations (1):
- Zelo Phase One Clinical Trial Unit, Bispebjerg Hospital, Copenhagen NV, Denmark

REFERENCES:
- [Background] Koppert W, Ihmsen H, Korber N, Wehrfritz A, Sittl R, Schmelz M, Schuttler J. Different profiles of buprenorphine-induced analgesia and antihyperalgesia in a human pain model. Pain. 2005 Nov;118(1-2):15-22. doi: 10.1016/j.pain.2005.06.030. Epub 2005 Sep 9. PMID 16154698
- [Result] Ravn P, Secher EL, Skram U, Therkildsen T, Christrup LL, Werner MU. Morphine- and buprenorphine-induced analgesia and antihyperalgesia in a human inflammatory pain model: a double-blind, randomized, placebo-controlled, five-arm crossover study. J Pain Res. 2013;6:23-38. doi: 10.2147/JPR.S36827. Epub 2013 Jan 9. PMID 23359655